CLINICAL TRIAL: NCT02172612
Title: Evaluation of a Patient-Centered Medication Therapy Management Intervention to Reduce Inappropriate Anticholinergic Prescribing in the Elderly
Brief Title: A Pilot Study to Reduce Inappropriate Anticholinergic Prescribing in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daniela Moga (Other)
Responsible Party: Sponsor-Investigator, Daniela Moga, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-0461-F3R
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Alzheimer Disease
Keywords: Anticholinergic drugs
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 - Intervention (Experimental): Those included in the intervention group will undergo an educational session with the study pharmacist and one of the licensed prescribers from Sanders-Brown to discuss recommended changes in their treatment plan. If changes in medications are indicated by the pharmacist-prescriber team, and accepted by the patient, new prescriptions will be provided and a letter will be sent to the primary care physicians detailing the changes made and the rationale behind such changes.
  Interventions: Other: Arm 1 Education Session
- Arm 2 - Control (No Intervention): Those included in the control group will receive a generic brochure about medication safety and inappropriate medication use in the elderly.

INTERVENTIONS:
Other: Arm 1 Education Session — Those included in the intervention group will undergo an educational session with the study pharmacist and one of the licensed prescribers from Sanders-Brown to discuss recommended changes in their treatment plan. If changes in medications are indicated by the pharmacist-prescriber team, and accepted by the patient, new prescriptions will be provided and a letter will be sent to the primary care physicians detailing the changes made and the rationale behind such changes.
  Arms: Arm 1 - Intervention

SUMMARY:
This will be an eight-week, prospective, placebo-controlled, randomized trial to evaluate a patient-centered team (pharmacist-physician) intervention to improve medication appropriateness and reduce the use of inappropriate anticholinergic medications in elderly patients enrolled in the Sanders-Brown Alzheimer's Disease Center (ADC) cohort.

DETAILED DESCRIPTION:
Screening: Patients seen in the Sanders-Brown clinic as part of the ADC cohort will be screened for eligibility in our study by the ADC study coordinator and the licensed prescriber involved in the scheduled ADC visit.

Enrollment: If the patient is considered eligible based on the screening, the study coordinator will introduce our study to the potential participant and will answer questions the patient might have. If the patient is interested, the study coordinator will obtain the informed consent and will proceed with the study related activities. Medication information and SF-36 are collected as part of the ADC cohort data collection; therefore, to reduce the burden on the participant, we are planning to work with the ADC team and use these data as baseline information for our study. For participants randomized to the intervention group, the two onsite study visits will be scheduled- the intervention visit will be planned within a week after enrollment and the end of study visit will be scheduled 8 weeks after enrollment. Participants randomized to the control group will have their end of study visit scheduled 8 weeks post-enrollment.

After enrollment, the study pharmacist will perform medication therapy management (MTM) to review all medications from the list provided by the patient. The pharmacist will identify any anticholinergic medication, will determine the medication appropriateness index and will prepare a report to include information on potential inappropriate medications to make recommendations for treatment discontinuation or change as considered appropriate. For participants included in the intervention group, the pharmacist will discuss the recommendations with one of the licensed prescribers before the scheduled visit by the participant. Final recommendations on discontinuing or changing inappropriate medications will be made by medical staff. In the case of medication necessity, safer alternatives will be sought and will be included in the proposed plan to be discussed with the patient assigned to the intervention arm.

Intervention visit: Those included in the intervention group will undergo an educational session with the study pharmacist and one of the licensed prescribers from Sanders-Brown to discuss recommended changes in their treatment plan. If changes in medications are indicated by the pharmacist-prescriber team, and accepted by the patient, new prescriptions will be provided and a letter will be sent to the primary care physicians detailing the changes made and the rationale behind such changes. Sending a letter to the primary care provider to inform of medication changes by the specialist is considered standard of care.

Both intervention and control group will receive a generic brochure that describes medication safety in the elderly in general terms.

End of study visit: At this visit, which will be scheduled eight weeks after enrollment, both the intervention and control group will complete SF-36 and will update the data on their current medication. They will also complete a questionnaire asking about their experience as part of the study.

Post-visit evaluation: The study pharmacist will review the new medication list and the follow-up MAI will be calculated through a similar procedure as detailed above.

Post-visit follow-up: All of the study participants will receive a thank you letter and will be informed of the availability of the study team to further discuss their medication plan and of the ADC prescribers to continue to support their ongoing care. The thank you letter will also include a check to compensate participants for being part of our study.

Intervention The intervention will be based on the pharmacist-physician team drug review. For patients randomized to the intervention group, the clinical pharmacist performed drug reviews will guide a revised medication plan that will be discussed with the patient. Specifically, the proposed plan will attempt to recommend discontinuation or replacement of any inappropriate drug with anticholinergic properties, with safer drug alternatives (i.e., with less or no anticholinergic activity). When drug alternatives are unavailable, reduction in dosage will be attempted to reduce the anticholinergic burden. As part of their routine clinical duties and care for ADC research participants, the prescribing team (ADC licensed practitioners) will make the recommendations to the patient, while the study pharmacist will be responsible for recommendations and provision of information to educate the patient about medication safety and the importance of patient involvement in medication awareness and oversight. Appropriate changes will be determined and carried out by the licensed prescriber and a letter will be sent informing the primary care physician of medication changes and rationale for such changes.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled at the Sander's Brown Center on Aging Alzheimer Disease Center
* Are 65 years of age or older
* Are taking at least one anticholinergic medication
* No cognitive impairment or mild cognitive impairment

Exclusion Criteria:

* Are younger than 65 years of age
* Have moderate to severe cognitive impairment
* Live in a long-term care facility

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-09; Primary Completion 2015-11-20 (Actual); Study Completion 2015-11-20 (Actual)

PRIMARY OUTCOMES:
Change in appropriateness of anticholinergic medication prescribing practices. | Two years
  This will be measured through the change in the appropriateness of anticholinergic medication prescribing from baseline to follow-up, as measured by the medication appropriateness index (MAI)

SECONDARY OUTCOMES:
Change in Anticholinergic Burden | 2 years
  The anticholinergic burden will be measured from baseline to follow-up, as measured by the anticholinergic drug scale (ADS).Anticholinergic burden (and change from baseline to follow-up) will be measure using the updated ADS score; the ADS has four levels for each included drug, ranging from 0 (no known anticholinergic activity) to 3 (markedly anticholinergic activity). The summation of anticholinergic activity level for all the drugs taken by a patient reflects the total anticholinergic burden.

OTHER OUTCOMES:
Change in perceived health status | 2 years
  Will be measured using the SF-36 at baseline and at the Week 8, End-of-study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela C Moga, MD, PhD, Principal Investigator — University of Kentucky
Locations (1):
- Sander's BrownCenter on Aging, Lexington, Kentucky, United States

REFERENCES:
- [Derived] Moga DC, Abner EL, Rigsby DN, Eckmann L, Huffmyer M, Murphy RR, Coy BB, Jicha GA. Optimizing medication appropriateness in older adults: a randomized clinical interventional trial to decrease anticholinergic burden. Alzheimers Res Ther. 2017 May 23;9(1):36. doi: 10.1186/s13195-017-0263-9. PMID 28535785